CLINICAL TRIAL: NCT04418869
Title: Metabolic Effects of Exercise in Adolescents With Type 1 Diabetes
Brief Title: Exercise in Adolescents With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 251981
Record Dates: First submitted 2020-05-15; First posted 2020-06-05 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Exercise; Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): All subject will perform three different exercise bouts and one control session.
  Interventions: Other: Exercise bouts

INTERVENTIONS:
Other: Exercise bouts — Each subject performed three bouts with 45 minutes of exercise (continuous exercise, intermittent exercise and resistance exercise) in a randomized order. In addition a control session were performed where the subjects sat on a chair for 45 minutes.

SUMMARY:
Regular physical activity is an important part of diabetes management in adolescents with type 1 diabetes (T1D). Increased physical activity has several beneficial effects such as improved lipid profile, insulin sensitivity and quality of life. In addition, a reduced HbA1c is often seen in association to increased physical activity. However, the effect on glycemic control and the acute glycemic response seems to differs between different types of exercise. This issue is poorly studied in adolescents with T1D and the mechanism behind this is not fully understood.

The primary aim of this study was to compare the acute effects on glycemia of resistance and two aerobic continuous and intermittent exercise bouts in adolescents with type 1 diabetes. Secondarily, the investigators want to compare the different exercise according to hormonal changes and expression of mRNA in muscle.

At a baseline visit the participants was tested for maximal oxygen consumption (pVO2peak) and maximal strength (1-RM). The study participants then performed three exercise bouts and one control session (resting), each on 45 minutes, in a randomized order. Measurement was performed during and after the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Type 1 diabetes
* HbA1c < 65 mol/mol at inclusion
* Regularly performing physical activity
* Aged 16-18 years old

Exclusion Criteria:

* Less than 0.5 U/kg in insulin requirements
* Duration of diabetes less than one year.

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Gender is based on personal identity number and self-identification.
Enrollment: 8 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in plasma glucose during exercise and recovery | Plasma glucose were measured at 5 minutes before and at start of the bouts. Thereafter glucose was measured at 5,10,15,30 and 45 minutes during exercise. In addition glucose were measured at 15, 30, 45 and 60 minutes during the initial recovery period.
  Plasma glucose (mmol/l) measured by an hand-held glucometer

SECONDARY OUTCOMES:
Sensor glucose | Blinded continuous glucose measurement was started when the exercise bouts were finished and were there after used during the next 22 hours (until the next morning at 08:00 am).
  Blinded continuous glucose measurement (mmol/l) were used to measure sensor glucose
Changes in levels of hormones during exercise and recovery | Serum samples were collected at baseline and after 15 ,30 ,45 of exercise and after 15 minutes of recovery for later analysis
  Insulin, glucagon, catecholamines, insulin-like growth factor I, cortisol, growth hormone
Change in levels of messenger ribonucleic acid (mRNA) between baseline and exercise. | One biopsy (baseline) were collected approximately one week before the first exercise bout and thereafter one biopsy appr. 60 minutes after each exercise bout.
  mRNA levels were analyzed with microarray from muscle biopsies and compared between exercise bouts and baseline.
Comparisons of levels of messenger ribonucleic acid (mRNA) between different exercise bouts. | One biopsy was collected appr. 60 minutes after each exercise bout.
  mRNA levels were analyzed with microarray from muscle biopsies and compared between the exercise bouts.
Change in heart rate during exercise. | Heart rate was monitored continuously during exercise from 5 minutes before start of exercise until the bout was finished (time-point 45 minutes).
  Heart rate (beats per minute) were monitored by pulse oximetry and compared between the exercise bouts.
Change in hemoglobin saturation during exercise. | Hemoglobin saturation was measured continuously during exercise from 5 minutes before start of exercise until the bout was finished (time-point 45 minutes).
  Hemoglobin saturation (SpO2 %) was monitored by pulse oximetry and compared between the exercise bouts.
Change in cardiac output. | Cardiac output was measured continuously during exercise from 5 minutes before start of exercise until the bout was finished (time-point 45 minutes).
  Cardiac output (L/min) was measured with Physioflow and compared between the exercise bouts.

CONTACTS AND LOCATIONS:
Overall Officials: Fawzi Kadi, Professor, Study Chair — School of health Sciences, Örebro University, Sweden

IPD SHARING:
Plan to Share IPD: No